CLINICAL TRIAL: NCT03242655
Title: Adaptation and Testing of a Primary Care HCV Group Medical Treatment Intervention
Brief Title: HCV Group Evaluation and Treatment Uptake (HCV GET-UP) Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6948; K23DA039060-03PD (NIH); K23DA039060-03 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis C; Substance Use Disorders
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Random Controlled Trials (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCV GET-UP (Group Intervention) (Experimental): HCV GET-Up (Group Evaluation and Treatment Uptake)
  Interventions: Behavioral: HCV GET-Up (Group Evaluation and Treatment Uptake)
- Control (No Intervention): Individual onsite HCV treatment at a primary care center

INTERVENTIONS:
Behavioral: HCV GET-Up (Group Evaluation and Treatment Uptake) — Groups will meet for 4 weekly 1-hour sessions facilitated by the PI and focused on providing education, motivation, and behavior change skills, along with an HCV medical evaluation. Patients will then be offered HCV treatment by individual provider after 4-week group evaluation and education intervention.
  Arms: HCV GET-UP (Group Intervention)

SUMMARY:
People who inject drugs (PWID) represent the overwhelming majority of both HCV and HIV/HCV infected people in the United States. Though new, direct-acting HCV medications are highly efficacious and have the potential to end the HCV epidemic, few PWIDs ever initiate treatment. This study seeks to improve HCV treatment uptake and cure among HCV and HIV/HCV+ PWIDs by testing a primary care based HCV Group Evaluation and Treatment UPtake (GET-UP) intervention. If efficacious, this innovative care intervention could provide a means to reduce the growing mortality from HCV, as well as decrease the current reservoir for HCV transmission.

DETAILED DESCRIPTION:
The goal of this proposal is to improve HCV (hepatitis C virus) treatment uptake among current and former injection drug users (IDUs) by testing an innovative, primary care based HCV Group Evaluation and Treatment UPtake (HCV GET-UP) intervention. IDUs make up the majority of the 4 million Americans chronically infected with HCV, and up to 90% of HIV+ IDUs are infected with HCV. In the U.S., HCV is the leading cause of end-stage liver disease and hepatocellular carcinoma, and the most common indication for liver transplantation. Without imminent action, mortality from HCV-related disease is projected to triple over the next decade and HCV-related deaths have already surpassed deaths related to HIV.

While past HCV therapies have been relatively ineffective, new oral treatment regimens with direct-acting antivirals are substantially more efficacious, with few side effects, and cure rates as high as 100% for both HCV+ and HIV/HCV+ individuals. Importantly, successful HCV treatment has been associated with decreased mortality. Unfortunately, there are significant gaps along the HCV care cascade that prevent patients from ever realizing the benefits of these revolutionary medications. Approximately 10% of all HCV+ patients, and even fewer IDUs, have ever initiated HCV treatment.

Given the ease and efficacy of the new HCV medications, investigators have an unprecedented opportunity to treat IDUs within medical settings that they are already accessing, such as primary care clinics. Community-based primary care clinics, such as Federally Qualified Health Centers (FQHCs), are abundant throughout the US and serve populations at high risk for HCV, such as IDUs; studies show an HCV prevalence rate of approximately 8% in FQHCs almost 5 times greater than the general population. Over the past year at Montefiore Medical Center, investigators have piloted onsite HCV treatment at one FQHC and treated nearly 50 patients (81% former or current IDUs) with direct-acting antivirals, with 93% cure rates.

Despite high HCV cure rates for those treated in primary care at our FQHC, only a small minority of eligible patients has initiated treatment. Though onsite treatment reduces obstacles related to specialty referral, patient level barriers to HCV evaluation and treatment uptake still exist. IDUs in particular often have limited HCV knowledge, as well as low perceived vulnerability to poor HCV-related health outcomes, low self-esteem and poor self-efficacy, high levels of perceived stigma, and mistrust of healthcare providers. These, as well as other barriers, prevent many IDUs from ever initiating HCV evaluation or starting the treatment uptake process. Investigators therefore propose to test an HCV Group Evaluation and Treatment UPtake (HCV GET-UP) intervention to improve HCV medical evaluation and treatment uptake for HCV and HCV/HIV IDUs within an FQHC. Group-based interventions, often familiar to IDUs, provide social support and encourage behavior change, which together promote enhanced engagement in care. Group-based care can also allow efficient delivery of health-education and medical treatment. Informed by the Information-Motivation-Behavior (IMB) model. Investigators hypothesize that a group-based HCV intervention, HCV GET-UP, delivered in an FQHC already accessed by patients, will improve HCV treatment uptake by: (1) providing HCV education; (2) increasing motivation by minimizing stigma, and addressing competing priorities and social norms; and (3) increasing self-efficacy and related behavioral skills. Investigator propose the following specific aims:

Aim 1: To assess the feasibility and acceptability of HCV GET-UP. Investigators will pre-test HCV GET-UP by conducting two group interventions (each consisting of 4 weekly sessions; 8 participants in each intervention group). Investigators will assess feasibility by examining process measures, and acceptability using a brief, self-administered questionnaire after each of the 4 sessions. Investigators will also conduct focus groups after the entire 4-session intervention. Investigators will then refine HCV GET-UP based on these findings.

Aim 2: To conduct a pilot randomized controlled trial of the efficacy of HCV GET-UP for improving HCV treatment uptake in an FQHC. Investigators will enroll 96 HCV+ or HIV/HCV+ IDUs and randomize them 1:1 to HCV GET-UP plus onsite treatment in primary care (intervention) versus onsite treatment alone (control). Our primary outcome is HCV treatment uptake, and secondary outcomes will include HCV medical evaluation, HCV treatment completion, and HCV cure.

Aim 3: To determine potential moderators and mediators of the impact of HCV GET-UP on HCV treatment uptake, using a sequential explanatory design. First, Investigators will perform exploratory quantitative analyses to determine if there are specific patient characteristics (demographic, clinical) that moderate the intervention effect, and if there are mediators (reduced stigma, peer support, increased self-efficacy) of HCV GET-UP's impact on treatment uptake. Second, investigators will perform semi-structured interviews with 20 participants randomized to HCV-GET UP to explore potential moderators/mediators deduced from quantitative analyses.

ELIGIBILITY:
Inclusion Criteria:

* HCV Ab+ with detectable HCV viral load
* greater than fifth grade reading level
* English proficiency
* current or former IDUs
* willingness to be randomized to a group intervention.

Exclusion Criteria:

* short life-expectancy, such that HCV treatment would not be beneficial (e.g. end-stage cancer)
* decompensated liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Hepatitis C Virus (HCV) Treatment Uptake | within 6 months after HCV medical Evaluation Visit
  First HCV medication prescription filled

SECONDARY OUTCOMES:
Hepatitis C Virus (HCV) medical evaluation | within 6 months after Baseline Research visit
  Sustained Virological Response at 12 weeks post-treatment (SVR12)
Hepatitis C Virus (HCV) treatment completion | 8 or 12 weeks depending on medication
  Completion will be tracked via pharmacy records
Hepatitis C Virus (HCV) cure | 12 weeks after treatment completion
  Sustained Undetectable HCV Viral Load at least 12 weeks post-treatment (SVR12)

CONTACTS AND LOCATIONS:
Overall Officials: Brianna L Norton, DO, MPH, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Comprehensive Health Care Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No